CLINICAL TRIAL: NCT04809103
Title: A Phase 1 Trial of Intratumoral Cisplatin for Early Stage, Resectable, Non-Small Cell Lung Cancer
Brief Title: Intratumoral Cisplatin for Resectable NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, C. Matthew Kinsey MD, MPH, Director, Interventional Pulmonary, University of Vermont
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 00001101
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intratumoral Cisplatin 20 mg (Experimental): Second dose level
  Interventions: Drug: cis-diamminedichloroplatinum
- Intratumoral Cisplatin 10 mg (Experimental): First dose level
  Interventions: Drug: cis-diamminedichloroplatinum

INTERVENTIONS:
Drug: cis-diamminedichloroplatinum — Cisplatin delivered bronchoscopically at the time of diagnosis of NSCLC
  Other Names: cisplatin

SUMMARY:
PRIMARY OBJECTIVE:

To identify the maximum tolerated dose (MTD) of intratumoral cisplatin, delivered during a single bronchoscopy with cone-beam CT confirmation, in a dose escalation protocol

DESIGN: 3+3 dose escalation.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is the leading cause of cancer-related death in the United States. Even for early stage disease, the rate of recurrence following surgical resection is as high as 50%. Although neoadjuvant therapy, administered before surgery, for early stage lung cancer is associated with a survival benefit, it is rarely used due to the systemic toxicity of intravenous (IV) cytotoxic chemotherapy. IV immunotherapies are also being evaluated in combination with systemic therapies in the neoadjuvant setting. However, only a minority of patients respond to immunotherapy. One of the most common reasons for failure of immunotherapy is lack of presentation of tumor antigens to the immune system, a problem that may be potentially addressed with cytotoxic agents.

Over the last several years, case series have demonstrated the feasibility and safety of delivering cisplatin directly into lung tumors. Given the current knowledge of safety and tolerability of intratumoral cisplatin, coupled with the potential to achieve immune priming that may help address systemic micrometastases, the investigators postulate that intratumoral cisplatin will be well-tolerated, and potentially effective, neoadjuvant therapy for patients with early stage, resectable, non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Eastern Cooperative Oncology Group performance status 0 or 1
* Patients must have adequate organ and marrow function as defined below:

  * Leukocytes ≥3,000/microliter
  * Platelets ≥100,000/microliter
  * Total bilirubin ≤ institutional upper limit of normal (ULN)
  * Aspartate aminotransferase /Alanine aminotransferase ≤3 × institutional upper limit of normal
  * Creatinine ≤ institutional ULN
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Have known or suspected clinical stage I-IIb NSCLC after computed tomography (CT) and/or positron emission tomography at time of enrollment
* Presence of a target lesion with a minimum volume of 1.0 cm3, (approximately1.2 cm in diameter) and ≤ 5.0 cm in diameter
* Agreement from a cardiothoracic surgeon, following review of past medical history, medications, pulmonary function testing, and CT scan that patient is likely to be a surgical candidate and that, after considering known possible adverse events, delivery of intratumoral cisplatin is unlikely to adversely affect surgical feasibility
* Rapid on-site cytopathologic examination (ROSE) performed during the procedure returns likely NSCLC (per the determination of a trained, attending, cytopathologist). No research procedures will be performed if ROSE is non-diagnostic
* A CT scan of the chest (with or without contrast) within 1 month of the screening visit
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Use of an investigational agent within 30 days of the screening visit
* IV chemotherapy within the 30 days of the screening visit
* Pregnancy/lactation (pregnancy test to be performed by pre-op as part of standard of care for women of child-bearing age as defined by University of Vermont Medical Center Policy
* History of prior radiation to the study lesion
* History of allergic reaction to cisplatin or its derivatives
* Patients with uncontrolled intercurrent illness
* Physician determination that patient would not be appropriate for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Matthew Kinsey, MD, MPH, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intratumoral Cisplatin 10 mg: First dose level in dose escalation study: Intratumoral cisplatin 10 mg.
  cis-diamminedichloroplatinum: Cisplatin delivered bronchoscopically at the time of diagnosis of NSCLC
- Intratumoral Cisplatin 20 mg: Second dose level in dose escalation study: Intratumoral cisplatin 20 mg.
  cis-diamminedichloroplatinum: Cisplatin delivered bronchoscopically at the time of diagnosis of NSCLC
Period: Overall Study
Arm/Group | Intratumoral Cisplatin 10 mg | Intratumoral Cisplatin 20 mg
Started | 3 (Consented) | 3
Completed | 3 (6 underwent delivery of intratumoral cisplatin as screening was ongoing during the procedure (diagnose, stage, and treat single procedure approach)) | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intratumoral Cisplatin 10 mg | Intratumoral Cisplatin 20 mg | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicity
Description: Adverse events as defined using the Common Terminology Criteria for Adverse Events
Time Frame: Within 2 weeks of delivery
Measure: Number; unit: participants
Groups:
- Intratumoral Cisplatin Arm: Single arm approach. There is no comparator or placebo group. Cisplatin will be administered directly into a non-small cell lung cancer, following imaging verification and pathologic diagnosis, during a single bronchoscopic procedure.
  cis-diamminedichloroplatinum: Cisplatin delivered bronchoscopically at the time of diagnosis of NSCLC
Arm/Group | Intratumoral Cisplatin Arm
Number analyzed (Participants) | 6
participants | 0

2. Secondary Outcome: Major Pathologic Response
Description: Evaluation of the tissue response to the drug
Time Frame: Assessed on the surgical resection specimen, performed within 30 days of bronchoscopic delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Intratumoral Cisplatin Arm
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: All possibly related Grade III CTCAE AEs were considered dose limiting
Arm/Group | Intratumoral Cisplatin 10 mg | Intratumoral Cisplatin 20 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intratumoral Cisplatin 10 mg (N=3) | Intratumoral Cisplatin 20 mg (N=3)
Headache (General disorders) | 0 (0) | 1 (1) — Patient developed headache 24h after the procedure, resolved with acetaminophen
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Developed non-productive cough with mild dyspnea 6 days after delivery. CXR without infiltrates, or evidence of pneumonitis. Resolved without treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04809103/Prot_SAP_000.pdf